CLINICAL TRIAL: NCT05745740
Title: An Open-label, Single-center, Phase Ib/II Study to Evaluate the Safety, Efficacy and Pharmacokinetics of RC48-ADC Combined With Pyrotinib in Local Advanced or Metastasis NSCLC With HER2 Mutation
Brief Title: A Study of RC48-ADC Combined With Pyrotinib For Treatment of Local Advanced or Metastasis NSCLC With HER2 Mutation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C021
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pyrotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48-ADC + Pyrotinib (Experimental)
  Interventions: Drug: RC48-ADC; Drug: Pyrotinib

INTERVENTIONS:
Drug: RC48-ADC — RC48-ADC 1.5/2.0 mg/kg by intravenous (IV) infusion, given on Day 1 of each 14-day cycle
  Other Names: DV
Drug: Pyrotinib — Pyrotinib 400 mg by oral once a day.

SUMMARY:
This study will evaluate the efficacy, safety and pharmacokinetics of RC48-ADC for injection combined with pyrotinib in subjects with local advanced or metastatic non-small cell lung cancer with HER2 mutation.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary agreement to provide written informed consent.
* Predicted survival ≥ 12 weeks.
* According to UICC/AJCC 8th Edition, histologically and/or cytologically-confirmed, cannot be surgically removed, locally advanced or metastatic NSCLC.
* Is willing and able to provide an adequate archival tumor tissue sample
* Has relapsed from or is refractory to standard treatment and had received both platinum-based therapy and immunotherapy.
* Measurable lesion according to RECIST 1.1.
* Documented HER2 exon 20 insertion mutation.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Adequate organ function.
* For female subjects: should be surgically sterilized, postmenopausal, or agree to use a medically approved contraceptive (such as an intrauterine device, contraceptives, or condoms) during study treatment and within 6 months after the end of study, the blood pregnancy test within 7 days of study enrollment must be negative and must be non-lactating. Male subjects: Patients who should be surgically sterilized or agree to use a medically approved contraceptive during the study treatment period and within 6 months after the end of the study.
* Willing and able to follow trial and follow-up procedures.

Exclusion Criteria:

* No known EGFR, ALK, ROS1, RET, NTRK, MET 14 or BRAF V600E mutation.
* Patient has had previous treatment with HER2-targeted therapy prior to study participation.
* History of major surgery within 4 weeks of planned start of trial treatment.
* Diagnosed with HBsAg, HBcAb positive and HBV DNA copy positive, or HCVAb positive, or HIVAb positive.
* Has received a live virus vaccine within 4 weeks of planned start of trial treatment.
* NYHA Class III heart failure.
* Suffering from active infection requiring systemic treatment.
* Uncontrolled hypertension, diabetes, Interstitial lung Disease, or COPD.
* Treated with systemic treatment (e.g. immunomodulators, corticosteroids or immunosuppressants) for the autoimmune disease within 2 years prior to the study treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
maximal tolerance dose (MTD) of RC48-ADC combined with Pyrotinib | DLT will be evaluated on 28 days of observation period
  Maximum-tolerated dose (MTD) was defined as the highest dose level at which no more than one of six patients experienced DLT during the DLT assessment window.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to approximately 3 years
  The objective response rate will be mainly analyzed by investigators according to the RECIST 1.1 standard tumor evaluation.
Disease control rate (DCR) | Up to approximately 3 years
  Disease control rate (DCR) is defined as cases where objective remission (assessed as complete remission or partial remission according to RECIST 1.1 standard) or stable disease during the study.
Duration of relief (DOR) | Up to approximately 3 years
  DOR is defined as the time from the first documented objective response (CR or PR) to the first documented disease progression or death.
Progression-free survival (PFS) | Up to approximately 3 years
  Progression-free survival (PFS) refers to the time from the date of randomization to the first researcher's evaluation of disease progression or death.
Overall survival (OS) | Up to approximately 3 years
  The objective response rate will be mainly analyzed by investigators according to the RECIST 1.1 standard tumor evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China